CLINICAL TRIAL: NCT06155877
Title: Interventions to Reduce Vaccine Hesitancy Among Adolescents: A Randomized Controlled Trial.
Brief Title: Testing The Effectiveness Of Two Interventions To Reduce Vaccine Hesitancy Among Adolescents
Acronym: Kidivax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National de la Recherche Scientifique, France (Other)
Collaborators: Université Paris-Dauphine (Unknown); Fondation La main à la pâte (Unknown); Direction de l Évaluation, de la Prospective et de la Performance (Unknown)
Responsible Party: Principal Investigator, Hugo Mercier, Research Director, Centre National de la Recherche Scientifique, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANR-21-SSMS-0006
Record Dates: First submitted 2023-11-09; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Vaccine Hesitancy; Vaccine Refusal; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Vaccination Hesitancy; Vaccination Refusal; Behavior

STUDY DESIGN:
Intervention Model Description: Participants were randomized at the school level, to minimize contamination between experimental conditions. Using administrative data, schools were stratified by their Priority Education status and by geographical categories (urban with high density, urban with medium density, rural). Then, within each stratum, schools were matched by triplets using the closest-neighbors approach, minimizing the quadratic distance between schools' success rate at the national end-of-middle school exam and Covid vaccination rate at the EPCI3 level. This resulted in 149 triplets. Within each triplet, schools were randomly assigned to one of the three experimental groups.
  Randomization code is available at the experiment's OSF repository:
  https://osf.io/rf5w9/?view_only=de759e4e36914c909adeac5fd541babf
Who Masked: Outcomes Assessor
Masking Description: For ethical reasons, pupils' parents were informed that their children would take part in an experiment aiming to test pedagogical materials about vaccination. Thus, the pupils were aware that they were participating in an experiment, and of the broad purpose of this experiment. However, the investigators asked teachers not to tell pupils about the different experimental conditions, and to arrange for another colleague to administer the questionnaires to their pupils. This limits the risk that pupils bias their behavior to fit the hypotheses associated with their experimental group - whether because of their own reaction or because of their teachers' reaction. Furthermore, since vaccination is part of the French national curriculum, the investigators argue that it is difficult for pupils to know whether the materials they were presented with is the standard one or one of our interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LAMAP intervention (Experimental): Teachers receive two sets of activities, accompanied by a tutorial. Both sets of activities also include evaluation tools that teachers can use to clarify the objectives of the lesson and to assess the pupils' learning progress. The estimated length of each set is 5 hours.The activities and the tutorials were created by pedagogical experts of the Fondation La Main à la pâte, an NGO whose goal is to foster science education. Activities and tutorials are now freely available on the La Main a la pâte website. Teachers were free to choose whether to present the first or the second set of activities, and to choose how many of the activities to conduct. The actual length of the intervention thus varied from one classroom to another, which mimics ecological conditions. Teachers were asked to devote at least one hour to the activities.
  LAMAP activities are available on the experiment's OSF repository
  Interventions: Behavioral: Activité Vaccins et Vaccination - LAMAP
- Chatbot intervention (Experimental): Teachers, and then pupils, receive a link to a chatbot. This chatbot is a basic conversational agent that can answer the most common questions about vaccination. The chatbot is entirely scripted, providing users with a limited choice of questions at each stage. These questions are the most commonly raised questions about vaccination in adolescents, based on existing literature, and on focus groups conducted by our team. In this intervention, teachers will be asked to supervise the use of the chatbot in class. Pupils will use the chatbot either individually or in groups depending on the number of computers available. Teachers will be encouraged to conclude the intervention by a class discussion. Teachers will be asked to devote about one hour to this intervention (use of the chatbot and class discussion). The full chatbot text is available on the experiment's OSF repository
  Interventions: Behavioral: Kidivax Chatbot
- Control (No Intervention): In the control group, teachers were not sent any extra materials, and pupils were exposed to the standard curriculum. Teachers in the control group received the material after the end of the intervention. French teachers most commonly offer the course on vaccination during the last year of middle school (the equivalent of 9th grade). Time spent on this course varies and can be quite small.

INTERVENTIONS:
Behavioral: Activité Vaccins et Vaccination - LAMAP — Two activities created by the La Main a la Pate foundation
  Arms: LAMAP intervention
Behavioral: Kidivax Chatbot — A chatbot created by our team to answer the most common questions about vaccination, based on a literature review and on focus groups.
  Arms: Chatbot intervention

SUMMARY:
Vaccines currently prevent several million deaths every year and more lives could be saved if vaccination take up increased. The World Health Organization identifies vaccine hesitancy as one of the ten most important threats to global health and emphasizes the importance of devising interventions to reduce vaccine hesitancy. The two most promising interventions rely on consensus messaging, which has robust but small effects, and interactive discussion, which has larger effects, but is difficult to scale up. School-based interventions aimed at adolescents have the potential to make the best of both types of interventions. Interventions that take place in schools can be conducted over longer periods of time (up to several hours) and are rolled out by a figure that is typically trusted and respected (the teacher). Moreover, intervening during adolescence is particularly timely since important vaccines are delivered at that age (most notably the human papillomavirus vaccine), and because attitudes towards vaccination during adolescence might have a long-lasting impact, as is the case for other health related attitudes.

This study tests the effectiveness of two interventions, a pedagogical intervention based on consensus messaging, and a chatbot intervention designed to mimic interactive discussion, on 9th grade French pupils.

ELIGIBILITY:
Inclusion Criteria:

* French 9th grade students (equivalent to "troisième")'
* One class per school

Exclusion Criteria:

* Do not understand French

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8590 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Attitude towards vaccination | Up to 8 months
  Participants' attitude towards vaccination were measured as the average agreement with 4 questions measured on a 7-points Likert Scale created for this study, ranging from 1 - "Completely disagree" to 7 - "Totally agree", where a higher score corresponds to more positive attitudes towards vaccination.
  "The vaccines used in France are effective" "The vaccines used in France are safe" "Vaccines are useful because they protect us from dangerous diseases". "It is important to get vaccinated to protect others". For the full questionnaire, see the experiment's OSF repository.
  All outcomes were assessed three times: before teachers received our interventions (November 15th - December 12th), in the middle of the school year (March 6th -June 8th), and after all teachers used our interventions (May 11th - June 23rd).

SECONDARY OUTCOMES:
Knowledge about vaccination | Up to 8 months
  Knowledge is measured as the average number of correct answers to 11 True or False questions:
  "Vaccines are not necessary, since diseases can be treated by drugs (such as antibiotics)" "Without vaccines, smallpox would still exist" "The effectiveness of vaccines has been scientifically proven" "Children would be more resistant if they did not receive so many vaccines" "Vaccination can cause certain disorders, such as autism, multiple sclerosis or diabetes" "If a child receives too many vaccines at once, it can overload their immune system" "The chemicals included in vaccines are not dangerous" "Vaccination increases the risk of developing allergies" "Vaccines are injected too early, which prevents children from building their immune systems" "Vaccines cannot cause the disease they protect against" "Thanks to scientific advances, scientists can create vaccines with fewer side effects"
  Like all other outcomes, knowledge was assessed three times during the year.
Intention to be vaccinated | Up to 8 months
  Intention to be vaccinated is measured as the average agreement with 5 questions, measured on a 7-points Likert Scale created for this study, ranging from 1 - "Completely disagree" to 7 - "Totally agree", where a higher score corresponds to a stronger intention to be vaccinated.
  "If a vaccine for a new disease becomes available, I would get vaccinated" "If an AIDS vaccine became available, I would get vaccinated" "If a common cold vaccine became available, I would get vaccinated" "If a gastroenteritis vaccine became available, I would get vaccinated" "If a vaccine for certain cancers became available, I would get vaccinated" For the full questionnaire, see the experiment's OSF repository
  All outcomes were assessed three times: before teachers received our interventions (November 15th - December 12th), in the middle of the school year (March 6th -June 8th), and after all teachers used our interventions (May 11th - June 23rd).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mercier, PhD, Principal Investigator — Institut Jean Nicod, Département d'études cognitives, École normale supérieure, Université PSL, EHESS, CNRS; Coralie Chevallier, PhD, Principal Investigator — Institut Jean Nicod, Département d'études cognitives, École normale supérieure, Université PSL, EHESS, CNRS
Locations (1):
- Institut Jean Nicod, Département d'études cognitives, École Normale Supérieure, Université PSL, EHESS, CNRS, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The chatbot discussion tree, as well as LAMAP activities, consent forms, questionnaires, randomization and analysis codes will be made available online on the OSF repository.
  All consenting participants' responses to the three questionnaires will be anonymized and made available online.
  Individual covariates obtained from the French ministry of education cannot be made available online, which includes parents' sociodemographics, participants' gender, age, and their results on the French national 6th grade entrance exam.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once the study is published, individual participant data and analysis scripts will be made available indefinitely at the study's OSF repository.
URL: https://osf.io/rf5w9

REFERENCES:
- See also: This experiment was pre-registered before data was collected on the OSF platform. This experiment is retroactively registered on an ICMJE-compatible database for publication needs. This is the final link for this repository, accessible after publication — https://osf.io/rf5w9
- See also: This experiment was pre-registered before data was collected on the OSF platform. This experiment is retroactively registered on an ICMJE-compatible database for publication needs. This is a temporary view-only link of this repository — https://osf.io/rf5w9/?view_only=de759e4e36914c909adeac5fd541babf